CLINICAL TRIAL: NCT01994512
Title: Swedish Spinal Stenosis Study. An RCT Comparing Decompression With Fusion to Decompression Only in Lumbar Spinal Stenosis With or Without Degenerative Olisthesis.
Brief Title: Swedish Spinal Stenosis Study
Acronym: SSSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS 01
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal stenosis; Decompression; Fusion; Olisthesis
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis | interventions — Decompression; Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decompression without fusion (Experimental): Surgery of the stenotic spinal segments with decompression of the neural elements without concommitant fusion.
  Interventions: Procedure: Decompression without fusion
- Decompression with fusion (Experimental): Surgery of the stenotic spinal segments with decompression of the neural elements with concommitant fusion.
  Interventions: Procedure: Decompression with fusion

INTERVENTIONS:
Procedure: Decompression without fusion — Decompressive surgery of both central and lateral component of the stenosis.
  Arms: Decompression without fusion
Procedure: Decompression with fusion — Decompressive surgery of both central and lateral component of the stenosis AND concomitant instrumented or uninstrumented posterior fusion of decompressed segments.
  Arms: Decompression with fusion

SUMMARY:
A national randomized multicentre trial (RCT) where decompression is compared with decompression with simultaneous fusion in 245 patients with spinal stenosis on one or two adjacent lumbar levels with or without degenerative olisthesis. The material is stratified for the existence of degenerative olisthesis >3mm. Monitoring is performed with clinical results from patient surveys after 2 and five years, and with radiological follow-up (MRI, CT and plain X-ray) and an objective function test (6 min walking test) after 2 years. The null hypothesis is that there is no difference in results between the two interventions.

ELIGIBILITY:
Inclusion Criteria:

* Pseudoclaudication in one or both legs and backpain (VAS>30)
* MRI with 1-2 adjacent stenotic segments (area <0.75 mm2)between L2 and sacrum
* Duration of symptoms >6 months
* Informed consent

Exclusion Criteria:

* Spondylolysis
* Degenerative lumbar scoliosis (Cobb angle >20 deg)
* History of lumbar spinal surgery for spinal stenosis or instability
* Stenosis not caused by degenerative changes
* Stenosis caused by herniated disc
* Other specific spinal conditions, Mb Bechterew, malignancy, neurologic disorders
* History of vertebral compression fractures in affected segments
* Psychological disorders where the surgeon considers participation inappropriate(dementia, drug abuse)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-10; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 2 years
  A difference in ODI of 12 at follow up between the two interventions is considered as significant.

SECONDARY OUTCOMES:
Back pain | 2 years
  The visual analog scale (VAS 0-100) is used the evaluate pain. A difference of 20 between the interventions is considered significant.
Leg pain | 2 years
  The visual analog scale (VAS 0-100) is used the evaluate pain. A difference of 20 between the interventions is considered significant.
EuroQol (EQ-5D) | 2 years
  Measurement of quality of life
Swiss Spinal Stenosis Questionnaire | 2 years
  A disease-specific self-report outcome instrument commonly used in trials to measure treatment outcomes in patients with lumbar spinal stenosis. The Swiss Spinal Stenosis Questionnaire quantifies severity of symptoms, physical function characteristics, and patient's satisfaction after treatment. It was designed to complement existing generic measures of lumbar spine disability and health status in the evaluation of patients with lumbar spinal stenosis.

REFERENCES:
- [Derived] Forsth P, Olafsson G, Carlsson T, Frost A, Borgstrom F, Fritzell P, Ohagen P, Michaelsson K, Sanden B. A Randomized, Controlled Trial of Fusion Surgery for Lumbar Spinal Stenosis. N Engl J Med. 2016 Apr 14;374(15):1413-23. doi: 10.1056/NEJMoa1513721. PMID 27074066